CLINICAL TRIAL: NCT01850498
Title: Motion Sensing Study in Epilepsy Patients
Brief Title: Epilepsy Motion Sensing
Status: Completed | Type: Observational
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Sponsor
Other Study IDs: 1663
Record Dates: First submitted 2012-11-01; First posted 2013-05-09 (Estimated); Last update posted 2013-05-09 (Estimated); Status verified 2013-05

CONDITIONS: Epilepsy
Keywords: Epilepsy; Seizure; Motor; Motion; Accelerometer
MeSH Terms: conditions — Epilepsy; Seizures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Partial seizures: Partial seizures with secondary generalization which results in visible clonic or tonic-clonic motor behavior
- Generalized seizures: Primarily generalized seizures (in patients with either primary [idiopathic] or secondary [symptomatic] generalized epilepsy), which may involve the following depending on the motor manifestation observed: myoclonic seizures, clonic seizures, tonic-clonic seizures, or atonic seizures.

SUMMARY:
Evaluate patient motion during seizures.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Diagnosed with epilepsy and expected to have at least one motor seizure in the EMU
* Determined by the Investigator to be an acceptable candidate for epilepsy evaluation with intracranial or scalp electrode monitoring
* Willing and able to wear 3 ActiGraph GT3X+ devices for the duration of their participation in the study and comply with the study protocol
* Have one of the following seizure types: (a) partial seizures with secondary generalization, which results in visible clonic or tonic-clonic motor behavior; (b) primarily generalized seizures (in patients with either primary [idiopathic] or secondary [symptomatic] generalized epilepsy), which may involve the following depending on the motor manifestation observed: myoclonic seizures, clonic seizures, tonic-clonic seizures, or atonic seizures.
* Be able to consent to participate by signing the Informed Consent document after a full explanation of the nature and purpose of this study
* Male or non-pregnant female
* English speaking

Exclusion Criteria:

* Currently enrolled in another investigational device, drug, or surgery study. Concurrent physiologic study participation is acceptable
* Have an implanted device that may interfere with GT3X+ recordings, ECoG/EEG recordings, ECG recordings, or video recordings
* Have a movement disorder that may affect GT3X+ recordings

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with epilepsy referred to epilepsy monitoring unit.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2012-05; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
To identify and evaluate seizure characteristics derived from an accelerometer that can be used in development of a seizure detection algorithm (compared to EEG readings). | While patients are being evaluated in an epilepsy monitoring unit.

SECONDARY OUTCOMES:
Evaluate the accuracy of an accelerometer in identifying seizures (compared to EEG readings). | While patients are being evaluated in an epilepsy monitoring unit.
Evaluate whether certain seizure types are more capable of being identified by the accelerometer (compared to EEG readings). | While patients are being evaluated in an epilepsy monitoring unit.
Evaluate heart rate and rhythm changes associated with seizure onset (compared to ECG readings). | While patients are being evaluated in an epilepsy monitoring unit.

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States